CLINICAL TRIAL: NCT04101721
Title: Randomized, Controlled, Multi-Center Study to Assess the Efficacy, Safety, and Tolerability of Intravitreal Aflibercept Compared to Laser Photocoagulation in Patients With Retinopathy of Prematurity
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of Intravitreal Aflibercept Compared to Laser Photocoagulation in Patients With Retinopathy of Prematurity
Acronym: BUTTERFLEYE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-ROP-1920; 2019-001764-29 (EudraCT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — aflibercept

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aflibercept Group (Experimental): Patients will receive a single intravitreal (IVT) injection per eligible eye at baseline.
  Interventions: Drug: aflibercept
- Laser Group (Experimental): Patients will undergo laser treatment in each eligible eye at baseline.
  Interventions: Procedure: laser photocoagulation

INTERVENTIONS:
Drug: aflibercept — Administered IVT
  Other Names: EYLEA®; REGN3; VEGF trap-eye; BAY86-5321
  Arms: Aflibercept Group
Procedure: laser photocoagulation — Transpupillary conventional laser will be administered according to standard local procedures.
  Arms: Laser Group

SUMMARY:
The primary objective of the study is to assess the efficacy of aflibercept compared to laser in patients diagnosed with retinopathy of prematurity (ROP). The secondary objectives of the study are to assess the need for a second treatment modality, to assess the recurrence of ROP in the study and to assess the safety and tolerability of aflibercept.

ELIGIBILITY:
Key Inclusion Criteria:

* Gestational age at birth ≤ 32 weeks or birth weight ≤1500 g
* Patients with treatment-naïve retinopathy of prematurity (ROP) classified according to the International Classification for ROP in at least one eye as:

  * Zone I Stage 1 plus, or 2 plus, or 3 non-plus or 3 plus, or
  * Zone II Stage 2 plus or 3 plus, or
  * Aggressive posterior retinopathy of prematurity (AP-ROP)

Key Exclusion Criteria:

* Known or suspected chromosomal abnormality, genetic disorder, or syndrome
* Previous exposure to any Intravitreal (IVT) or systemic anti-vascular endothelial growth factor (VEGF) agent, including maternal exposure during pregnancy and/or during breastfeeding
* Clinically significant neurological disease (eg, intraventricular hemorrhage grade 3 or higher, periventricular leukomalacia, congenital brain lesions significantly impairing optic nerve function, severe hydrocephalus with significantly increased intracranial pressure)
* Pediatric conditions rendering the infant ineligible for study intervention at baseline or for repeated blood draws as evaluated by a neonatal intensive care unit specialist and a study ophthalmologist
* Presence of active ocular infection within 5 days of the first treatment
* Advanced stages of ROP with partial or complete retinal detachment (ROP stage 4 and stage 5)
* ROP involving only Zone III

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (46):
- United States (24):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, La Jolla, California
  - Regeneron Study Site, Loma Linda, California
  - Regeneron Study Site, Orange, California
  - Regeneron Study Site, Palo Alto, California
  - Regeneron Study Site, San Diego, California
  - Regeneron Study Site, San Francisco, California
  - Regeneron Study Site, Gainesville, Florida
  - Regeneron Study Site, Augusta, Georgia
  - Regeneron Study Site, Chicago, Illinois
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Royal Oak, Michigan
  - Regeneron Study Site, Brooklyn, New York
  - Regeneron Study Site, Buffalo, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Valhalla, New York
  - Regeneron Study Site, Cleveland, Ohio
  - Regeneron Study Site, Oklahoma City, Oklahoma
  - Regeneron Study Site, Providence, Rhode Island
  - Regeneron Study Site, Austin, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Morgantown, West Virginia
- Bulgaria (2):
  - Regeneron Study Site, Sofia
  - Regeneron Study Site, Varna
- Colombia (2):
  - Regeneron Study Site, Medellín, Antioquia
  - Regeneron Study Site, Floridablanca, Santander Department
- Regeneron Study Site, Ostrava-Poruba, Czechia
- Regeneron Study Site, Debrecen, Hungary
- Regeneron Study Site, Iași, Romania
- Russia (2):
  - Regeneron Study Site, Saint Petersburg, Sankt-Peterburg
  - Regeneron Study Site, Moscow
- Regeneron Study Site, Bratislava, Slovakia
- Regeneron Study Site, Cheonan, South Korea
- Regeneron Study Site, Kaohsiung City, Taiwan
- Thailand (5):
  - Regeneron Study Site, Pathum Wan, Bangkok
  - Regeneron Study Site, Ratchathewi, Bangkok
  - Regeneron Study Site, Hat Yai, Changwat Songkhla
  - Regeneron Study Site, Chiang Mai, Chiang Mai
  - Regeneron Study Site, Khon Kaen
- Turkey (Türkiye) (3):
  - Regeneron Study Site, Adana
  - Regeneron Study Site, Ankara
  - Regeneron Study Site, Eskişehir
- Vietnam (2):
  - Regeneron Study Site, Ho Chi Minh City
  - Regeneron Study Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 137 participants were screened, 127 were randomized.
Pre-assignment Details: Of the 127 participants randomized, 33 were randomized to laser and 94 were randomized to aflibercept. Six of the 33 participants randomized to laser were withdrawn before receiving any study intervention (5 due to Parent/Guardian and 1 due to Physician decision); One of the 94 participants randomized to aflibercept was withdrawn before receiving any study intervention due to Parent/Guardian. In total, 120 participants (27, laser group; 93, aflibercept group) received at least 1 study treatment.
Units Other Than Participants: Eyes
Groups:
- Laser Photocoagulation: Participants received laser treatment to each eligible eye at baseline (Day 1), with supplementary laser treatments allowed. Multiple sessions within one week from baseline were counted as a single treatment. If both eyes were eligible, they were assigned to the same treatment group.
- Aflibercept 0.4 mg: Participants received one intravitreal injection of aflibercept 0.4 mg (0.01 mL) per eligible eye at baseline (Day 1), with up to 2 re-injections at the same single dose allowed for each eligible eye if required and interval since last aflibercept injection was 28 or more days. If both eyes were eligible, they were assigned to the same treatment group.
Period: Overall Study
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Started (Randomized and Treated) | 27; 50 Eyes | 93; 179 Eyes
Completed | 26; 48 Eyes | 87; 168 Eyes
Not Completed | 1; 2 Eyes | 6; 11 Eyes
Not completed — Withdrawal By Parent/Guardian | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized participants who received any study treatment. Eyes analyzed includes all treated eyes.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg | Total
Number analyzed (Participants) | 27 | 93 | 120
Number analyzed (Eyes) | 50 | 179 | 229
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Chronological Age at Randomization (date of randomization - date of birth + 1)
  Weeks | 11.09 (4.338) | 9.76 (3.149) | 10.06 (3.476)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 52 | 62
  Male | 17 | 41 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 16 | 20
  Not Hispanic or Latino | 22 | 72 | 94
  Unknown or Not Reported | 1 | 5 | 6
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 11 | 26 | 37
    Black or African American | 2 | 6 | 8
    Asian | 13 | 44 | 57
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 1 | 12 | 13
    Not Reported | 0 | 5 | 5
Retinopathy of prematurity (ROP) Zone, by eye [Count of Units; unit: Eyes] — ROP was classified by the investigator according to the International Classification for ROP in at least 1 eye with 1 of the following retinal findings: Zone I, or Zone II, or AP(aggressive posterior)-ROP (Zone I, Zone II). Zone I is the innermost zone of the retina centered around the optic disc, surrounded by the more peripheral Zone II. AP-ROP is a rapidly progressive form of ROP, with posterior location, commonly observed in Zone I, less common in posterior Zone II. AP-ROP, if untreated, usually progresses to retinal detachment. Eyes with AP-ROP are not always exclusive of disease stage.
  Eyes
    Zone I | 13 | 47 | 60
    Zone II | 37 | 132 | 169

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Absence of Active Retinopathy of Prematurity (ROP) and Unfavorable Structural Outcomes From Baseline to Week 52 of Chronological Age
Description: Active ROP was ROP requiring treatment and unfavorable structural outcome was defined as retinal detachment, macular dragging, macular fold, or retrolental opacity. For participants with both eyes enrolled in the study, both eyes must have met the endpoint. Participants with only one study eye enrolled were responders if the respective eye responded.
Time Frame: Baseline to week 52 of chronological age
Population: Full analysis set (FAS): All randomized participants who received any study treatment. Analysis on the FAS was performed according to the treatment assigned at baseline (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Number analyzed (Participants) | 27 | 93
Percentage of participants | 77.8 | 79.6
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Aflibercept 0.4 mg; Difference with confidence interval (CI) is calculated using Mantel-Haenszel weighting scheme adjusted by baseline ROP status; Test type: Non-Inferiority — Non-inferiority margin is 5%; Adjusted difference = 1.81, 95.1% CI 2-sided [-15.71 to 19.33]

2. Secondary Outcome: Percentage of Participants Requiring Intervention With a Second Treatment Modality From Baseline to Week 52 of Chronological Age
Description: Second treatment modality includes any treatment in addition to that assigned to the participant at baseline. This includes per-protocol rescue treatment (laser for aflibercept group, aflibercept for laser group), anti-VEGF agents not part of study protocol (e.g., bevacizumab, ranibizumab, commercially-available aflibercept not provided as study medication), or any ocular surgery for the management of any retinal pathology secondary to ROP (e.g., victrectomy, scleral buckle for retinal detachments).
Time Frame: Baseline to to week 52 of chronological age
Population: Full analysis set (FAS): All randomized participants who received any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Number analyzed (Participants) | 27 | 93
Percentage of participants | 18.5 | 15.1
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Aflibercept 0.4 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Adjusted difference = -3.66, 95.1% CI 2-sided [-19.86 to 12.54]

3. Secondary Outcome: Percentage of Participants With Recurrence of ROP Through Week 52 of Chronological Age
Description: Recurrence of disease is defined as the reappearance of the disease requiring further treatment (including retreatment or rescue), where both "presence of ROP" and "presence of active ROP requiring treatment" are marked as "Yes", after initial regression. Here, the initial regression is defined as, at a particular visit, absence of ROP or ROP treatment not required for active ROP, i.e., presence of ROP is marked as "No" or the presence of active ROP requiring treatment is marked as "No."
Time Frame: Baseline to week 52 of chronological age
Population: Full analysis set (FAS): All randomized participants who received any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Number analyzed (Participants) | 27 | 93
Percentage of participants | 29.6 | 39.8
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Aflibercept 0.4 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Adjusted difference = 10.10, 95.1% CI 2-sided [-9.83 to 30.02]

4. Secondary Outcome: Percentage of Participants With Ocular Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Time Frame: Baseline to Week 52 of chronological age
Population: Safety analysis set (SAF): All randomized participants who received any study treatment (active or laser); it is based on the treatment actually received (as treated).
Measure: Number; unit: Percentage of participants
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Number analyzed (Participants) | 27 | 93
Percentage of participants
  % Ocular TEAEs | 25.9 | 18.3
  % Ocular TESAEs | 11.1 | 6.5

5. Secondary Outcome: Percentage of Participants With Systematic (Non-ocular) TEAEs and TESAEs
Time Frame: Baseline to Week 52 of chronological age
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
Number analyzed (Participants) | 27 | 93
Percentage of participants
  % Systematic TEAEs | 51.9 | 47.3
  % Systematic TESAEs | 7.4 | 12.9

ADVERSE EVENTS:
Time Frame: From signing of informed consent form (ICF) to end of study (week 52 of chronological age visit), an average of 42 weeks
Description: Thirty-three (33) participants were randomized to laser and 94 participants randomized to aflibercept; however, 6 laser participants and 1 aflibercept participant were not treated and therefore, excluded from the safety analysis set (SAF) and FAS. SAF and FAS populations are identical: 27 laser group; 93 aflibercept group.
Arm/Group | Laser Photocoagulation | Aflibercept 0.4 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/93
Serious Adverse Events (participants affected / at risk) | 12/27 | 32/93
Other Adverse Events (participants affected / at risk) | 12/27 | 40/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser Photocoagulation (N=27) | Aflibercept 0.4 mg (N=93)
Bronchiolitis (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Poor feeding infant (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Overfeeding of infant (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Prophylaxis against dehydration (Surgical and medical procedures) | 0 (0) | 1 (1)
Removal of foreign body from gastrointestinal tract (Surgical and medical procedures) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Retinal detachment Study Eye (Eye disorders) | 2 (3) | 6 (7)
Vitreous haemorrhage Study Eye (Eye disorders) | 0 (0) | 2 (2)
Atrophy of globe Study Eye (Eye disorders) | 0 (0) | 1 (1)
Maculopathy Study Eye (Eye disorders) | 0 (0) | 1 (1)
Corneal infiltrates Study Eye (Eye disorders) | 1 (1) | 0 (0)
Retinal scar Study Eye (Eye disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser Photocoagulation (N=27) | Aflibercept 0.4 mg (N=93)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 4 (6)
Bacterial disease carrier (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 6 (7)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (8)
Conjunctival haemorrhage Study Eye (Eye disorders) | 0 (0) | 5 (7)
Strabismus Study Eye (Eye disorders) | 0 (0) | 6 (9)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04101721/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT04101721/SAP_003.pdf